CLINICAL TRIAL: NCT03466749
Title: A Real-world Study in China: the Safety and Efficacy of Paclitaxel Eluting Balloon Catheter in Coronary De-novo Lesions Treatment
Brief Title: Paclitaxel Eluting Balloon Catheter in Coronary De-novo Lesions Treatment in China
Acronym: RESPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Hospital of Jilin University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Tang-Du Hospital (Other); China-Japan Union Hospital, Jilin University (Other); Xuzhou Third People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, Doctor, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20172081
Record Dates: First submitted 2018-02-05; First posted 2018-03-15 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Drug eluting balloon; De-novo lesions
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Paclitaxel Eluting Balloon Catheter treatment
  Interventions: Device: Paclitaxel Eluting Balloon Catheter

INTERVENTIONS:
Device: Paclitaxel Eluting Balloon Catheter — Paclitaxel Eluting Balloon Catheter

SUMMARY:
The aim of this Real-world study in China is evaluating the Safety and Efficacy of Paclitaxel Eluting Balloon Catheter in Coronary de-novo lesions(target vessel diameter:2.5mm-4.0mm)Treatment. And the primary point of this study is the target lesion failure of 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-78 years of age, male or non-pregnant female;
2. patients with asymptomatic or symptomatic myocardial ischemia, stable or unstable angina pectoris, myocardial infarction with a course of more than two weeks, and patients with indications for percutaneous coronary intervention;
3. the target lesions were primary, in situ coronary artery stenosis, located on one or two different coronary artery vessels, the number of target lesions on each coronary artery was not more than one;
4. the length of the target lesion ≤ 26mm (visual), which can be covered by a single drug balloon (it is suggested that the balloon should cover at least 4mm healthy partition, 2 mm at each end; The reference diameter of target vessel was 2.5mm-4.0mm (visual);
5. the stenosis degree of the target lesion was ≥ 70%;
6. left ventricular ejection fraction ≥ 45%.
7. patients who can understand the purpose of the trial, voluntarily participate and sign informed consent, and are willing to follow up the study.

Exclusion Criteria:

Related to patients:

1. patients with myocardial infarction within two weeks;
2. pregnant or lactating women;
3. cardiogenic shock, acute infection, known bleeding or coagulation disorder, or active digestive tract; Patients with history of hemorrhage or ulcer, cerebral hemorrhage or subarachnoid hemorrhage, stroke within half a year;
4. patients with a life expectancy less than one year or with difficulties in clinical follow-up;
5. patients who had a history of PTCA or had other operations scheduled during the follow-up period of one year;
6. patients who are participating in any other clinical study and who have not reached the main end point of the study;
7. present or previous history of severe liver disease, and / or renal impairment: serum creatinine > 2.0 mg / dl( 176.8 umol / L) or undergoing hemodialysis therapy. Therefore, it does not meet the requirements of angiography;
8. patients with left ventricular ejection fraction below 45%;
9. for other reasons, the researchers did not think it was appropriate for a patient to be selected.

Related to lesions:

1. left main lesion and the bifurcation with side branch >2.5 mm;
2. the location of the lesion was less than 10 mm at the proximal end of the anterior descending branch, 5 mm in the circumflex branch and 5 mm in the proximal end of the right coronary artery.
3. severe calcification and twisted lesions which can not be successfully predilated, are not suitable for drug balloon delivery and expansion.
4. lesion length ≥ 26 mm;
5. evidence of severe thrombosis in target vessels before intervention;
6. lesions that cannot be treated with PTCA or other interventional techniques;
7. after predilation of the target lesion, residual stenosis ≥ 30% or TIMI blood flow < 3, and / or obvious flow limiting dissection.

Exclusion criteria related to drugs:

1. patients with bleeding constitution, anticoagulant or antiplatelet drugs;
2. patients who cannot tolerate aspirin and / or clopidogrel or who have a history of neutropenia or thrombocytopenia or who have too severe liver failure to receive clopidogrel;
3. patients known to be intolerant or allergic to heparin, contrast agents, paclitaxel, iopramide, rapamycin, polylactic acid-glycolic acid polymer, stainless steel, etc.
4. leukopenia (leukocyte count < 3 × 109 / L and the course > 3 days) or neutropenia ANC < 1000 neutrophil / mm3 and the course> 3 days). Or patients had a history of thrombocytopenia (< 100,000 platelets / mm3;
5. patients with a history of peptic ulcer or gastrointestinal bleeding in the past 6 months.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-02-22 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
TVF of 12 months after surgery | 12 months after surgery
  target vessel failure of 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, Ph.D.,M.D., Principal Investigator — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Undecided